CLINICAL TRIAL: NCT05786638
Title: Efficacy of Sublingual Versus Subcutaneous Allergen Immunotherapy in Patients With Bronchial Asthma
Acronym: Sublingual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Assistant lecturer, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD.21.09.522.R1
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Efficacy, Self
Keywords: Sublingual; subcutaneous; allergen immunotherapy
MeSH Terms: interventions — Desensitization, Immunologic

STUDY DESIGN:
Intervention Model Description: Sublingual versus subcutaneous allergen immunotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sublingual immunotherapy (Active Comparator): 50 Bronchial asthma (BA) patients received Sublingual immunotherapy
  Interventions: Drug: Allergen Immunotherapy Extract
- Subcutaneous immunotherapy (Active Comparator): 50 BA patients received Subcutaneous immunotherapy
  Interventions: Drug: Allergen Immunotherapy Extract

INTERVENTIONS:
Drug: Allergen Immunotherapy Extract — Sublingual subcutaneous allergen immunotherapy

SUMMARY:
Asthma is characterized by airway inflammation and is manifested by acute episodes of obstruction related to loss of control of airway inflammation mostly in response to a viral respiratory tract infection .The significance of eosinophilic inflammation in asthma is well established.

Late clinical reactions in asthma are associated with increase of immunoglobulin E (IgE) in serum. Serum IgE can be used as a measure of allergen provocation causing increased eosinophil activity. Serum IgE can be used to assess the exposure to environmental allergens, or decreasing presence of allergen in the environment and the need for increase or reduction of therapy.

Allergen immunotherapy is defined as the repeated administration of specific allergens to patients with IgE-mediated conditions for the purpose of providing protection against the allergic symptoms and inflammatory reactions associated with natural exposure to these allergens.

The aim of this work is to evaluate the effect of sublingual versus subcutaneous allergen immunotherapy as regard clinical response, serum IgE and sputum eosinophils

DETAILED DESCRIPTION:
study was conducted in Mansoura University Hospitals, Chest Medicine Department on patients attended to Asthma and Allergy clinic. The asthma symptoms and leukotrienes antagonist, inhaled B2 agonist, inhaled steroid and systemic steroid usage recorded throughout the study period. Venous blood and sputum samples were collected before and at the end of the study for determination of IgE and sputum eosinophil levels respectively. Fifty asthmatic patients recruited from Mansoura university allergy outpatient clinic were included before treatment with subcutaneous immunotherapy (SCIT) vaccines and another Fifty asthmatic patients were included before treatment with sublingual immunotherapy (SLIT) vaccines. In this study, All of patients were symptomatic and on medications either bronchodilators or inhaled corticosteroids (ICS). All patients were diagnosed by previous pulmonary function test (PFT) with reversibility test and follow up with our outpatient clinic (OPC). Each patient underwent spirometry to determine forced expiratory volume at 1st second (FEV1) and to ensure that his condition is stable before starting immunotherapy. Serum IgE and sputum eosinophil count were measured in 100 patients with asthma before and after 6 , 12 , 18 months of treatment with immunotherapy vaccines.

ELIGIBILITY:
Inclusion Criteria:

* New cases of allergic asthma indicated for immunotherapy (partially controlled by medical treatment with frequent exacerbations)
* Age >18 years

Exclusion Criteria:

* Pregnancy
* Co morbidity such as diabetes, hypertension, ischemic heart, malignancy
* Other causes of the increase in eosinophil as: parasitic infestation
* Acute exacerbation of BA
* Smoker
* Severe persistent asthma

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Total Ig E | After 6 month
  Measure Total igE after 6 months post immunotherapy
Total Ig E | After 12 month
  Measure Total igE after 12 months post immunotherapy
Total Ig E | After18 month
  Measure Total igE after 18 months post immunotherapy
Sputum eosinophil | After 6 month
  Measure Sputum eosinophil after 6 months post immunotherapy
Sputum eosinophil | After 12 month
  Measure Sputum eosinophil after 12 months post immunotherapy
Sputum eosinophil | After 18 month
  Measure Sputum eosinophil after 18 months post immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Elmoniem, Principal Investigator — Mansoura university Faculty of medicine
Locations (1):
- Mansoura university Faculty of medicine, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eifan AO, Akkoc T, Yildiz A, Keles S, Ozdemir C, Bahceciler NN, Barlan IB. Clinical efficacy and immunological mechanisms of sublingual and subcutaneous immunotherapy in asthmatic/rhinitis children sensitized to house dust mite: an open randomized controlled trial. Clin Exp Allergy. 2010 Jun;40(6):922-32. doi: 10.1111/j.1365-2222.2009.03448.x. Epub 2010 Jan 20. PMID 20100188
- [Result] Calderon MA, Demoly P, Casale T, Akdis CA, Bachert C, Bewick M, Bilo BM, Bohle B, Bonini S, Bush A, Caimmi DP, Canonica GW, Cardona V, Chiriac AM, Cox L, Custovic A, De Blay F, Devillier P, Didier A, Di Lorenzo G, Du Toit G, Durham SR, Eng P, Fiocchi A, Fox AT, van Wijk RG, Gomez RM, Haathela T, Halken S, Hellings PW, Jacobsen L, Just J, Tanno LK, Kleine-Tebbe J, Klimek L, Knol EF, Kuna P, Larenas-Linnemann DE, Linneberg A, Matricardi M, Malling HJ, Moesges R, Mullol J, Muraro A, Papadopoulos N, Passalacqua G, Pastorello E, Pfaar O, Price D, Del Rio PR, Rueff R, Samolinski B, Scadding GK, Senti G, Shamji MH, Sheikh A, Sisul JC, Sole D, Sturm GJ, Tabar A, Van Ree R, Ventura MT, Vidal C, Varga EM, Worm M, Zuberbier T, Bousquet J. Allergy immunotherapy across the life cycle to promote active and healthy ageing: from research to policies: An AIRWAYS Integrated Care Pathways (ICPs) programme item (Action Plan B3 of the European Innovation Partnership on active and healthy ageing) and the Global Alliance against Chronic Respiratory Diseases (GARD), a World Health Organization GARD research demonstration project. Clin Transl Allergy. 2016 Nov 23;6:41. doi: 10.1186/s13601-016-0131-x. eCollection 2016. PMID 27895895
- [Result] Fan TC, Chang HT, Chen IW, Wang HY, Chang MD. A heparan sulfate-facilitated and raft-dependent macropinocytosis of eosinophil cationic protein. Traffic. 2007 Dec;8(12):1778-1795. doi: 10.1111/j.1600-0854.2007.00650.x. Epub 2007 Oct 15. PMID 17944807
- [Result] Kundig TM, Bachmann MF. Allergen-specific immunotherapy: regulatory T cells or allergen-specific IgG? Hum Vaccin. 2010 Aug;6(8):673-5. doi: 10.4161/hv.6.8.12007. No abstract available. PMID 20523122
- [Result] Trautmann A, Schmid-Grendelmeier P, Kruger K, Crameri R, Akdis M, Akkaya A, Brocker EB, Blaser K, Akdis CA. T cells and eosinophils cooperate in the induction of bronchial epithelial cell apoptosis in asthma. J Allergy Clin Immunol. 2002 Feb;109(2):329-37. doi: 10.1067/mai.2002.121460. PMID 11842305